CLINICAL TRIAL: NCT05464693
Title: Clinical-Microbiological Evaluation of the Obstructive Biliary Disease
Brief Title: Microbiology in Obstructive BIliary Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. med. Hector Eloy Tamez Perez, Clinical professor, Hospital Universitario Dr. Jose E. Gonzalez
Other Study IDs: GA21-00003
Record Dates: First submitted 2022-06-15; First posted 2022-07-19 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Biliary Disease
MeSH Terms: conditions — Gallbladder Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with obstructive biliary disease: Patients admitted to hospital due to obstructive biliary disease secondary to benign and malign etiologies, undergoing ERCP, will be selected. Bile sample will be taken in ERCP procedure with sterile technique. Its macroscopic appearance will be assessed and biliary culture will be performed.
  Interventions: Diagnostic Test: ERCP biliary culture

INTERVENTIONS:
Diagnostic Test: ERCP biliary culture — The sample of biliary aspirate will be assessed as follows.
  1. Its macroscopic appearance will be analyzed: yellow, black, or purulent.
  2. Biliary culture will be performed; if bacterial growth is observed, its identification will be carried out by means of MALDI-TOF MS mass spectrometry and antibiotic susceptibility tests will be carried out, using the automated VITEK system.
  Other Names: MALDI-TOF MS mass spectrometry for bacteria identification; Antibiotic susceptibility for identified bacteria

SUMMARY:
Patients admitted to hospital due to obstructive biliary disease secondary to benign and malign etiologies, undergoing ERCP, will be selected. Bile sample will be taken in ERCP procedure with sterile technique. Its macroscopic appearance will be assessed and biliary culture will be performed.

DETAILED DESCRIPTION:
The sample of biliary aspirate will be assessed as follows.

1. Its macroscopic appearance will be analyzed: yellow, black, or purulent.
2. Biliary culture will be performed; if bacterial growth is observed, its identification will be carried out by means of MALDI-TOF MS mass spectrometry and antibiotic susceptibility tests will be carried out, using the automated VITEK system.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis or suspicion of biliary obstruction of any cause
* Any gender
* Over 18 years of age

Exclusion Criteria:

* Patients referred and previously treated at another hospital/clinic
* Previous ERCP
* Pregnancy
* Patient refusal to enter the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Emergency Department with a diagnosis of obstructive biliary disease of any cause, according to clinical, laboratory, and imaging data, who have indicated an Endoscopic Retrograde Cholangiopancreatography as part of their management.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of bacterial isolation in the obstructive biliary disease measured by percentage calculation | 1 year
  Determine the prevalence by percentage measurement of bacterial isolation in bile fluid in the obstructive biliary disease in patients undergoing ERCP.

SECONDARY OUTCOMES:
Bacteria in the obstructed bile duct | 1 year
  Isolate and identify most common bacteria that colonize and infect the obstructed bile duct by means of biliary culture and MALDI-TOF MS mass spectrometry, respectively
Antibiotic susceptibility of isolated bacteria in bile fluid | 1 year
  Determine antibiotic susceptibility of the isolated bacteria in bile fluid of patients with obstructed bile duct by means of the automated VITEK system
Bacteria and etiology of obstructive biliary disease | 1 year
  Association between isolated bacteria and the etiology of obstructive biliary disease

CONTACTS AND LOCATIONS:
Overall Officials: Joel Omar Jáquez Quintana, Principal Investigator — Hospital Universitario Dr. Jose E. Gonzalez
Locations (1):
- Marusia González Villarreal, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No
No data sharing plan

REFERENCES:
- [Background] European Association for the Study of the Liver (EASL). Electronic address: easloffice@easloffice.eu. EASL Clinical Practice Guidelines on the prevention, diagnosis and treatment of gallstones. J Hepatol. 2016 Jul;65(1):146-181. doi: 10.1016/j.jhep.2016.03.005. Epub 2016 Apr 13. No abstract available. PMID 27085810
- [Background] Bornman PC, van Beljon JI, Krige JE. Management of cholangitis. J Hepatobiliary Pancreat Surg. 2003;10(6):406-14. doi: 10.1007/s00534-002-0710-1. PMID 14714159
- [Background] Ehrenstein BP, Salamon L, Linde HJ, Messmann H, Scholmerich J, Gluck T. Clinical determinants for the recovery of fungal and mezlocillin-resistant pathogens from bile specimens. Clin Infect Dis. 2002 Apr 1;34(7):902-8. doi: 10.1086/339209. Epub 2002 Feb 26. PMID 11880954
- [Background] Kwon JS, Han J, Kim TW, Oh JH, Kwon HH, Jung JT, Kwon JG, Kim EY, Kim HG. Changes in causative pathogens of acute cholangitis and their antimicrobial susceptibility over a period of 6 years. Korean J Gastroenterol. 2014 May;63(5):299-307. doi: 10.4166/kjg.2014.63.5.299. PMID 24870302
- [Background] Gomi H, Solomkin JS, Schlossberg D, Okamoto K, Takada T, Strasberg SM, Ukai T, Endo I, Iwashita Y, Hibi T, Pitt HA, Matsunaga N, Takamori Y, Umezawa A, Asai K, Suzuki K, Han HS, Hwang TL, Mori Y, Yoon YS, Huang WS, Belli G, Dervenis C, Yokoe M, Kiriyama S, Itoi T, Jagannath P, Garden OJ, Miura F, de Santibanes E, Shikata S, Noguchi Y, Wada K, Honda G, Supe AN, Yoshida M, Mayumi T, Gouma DJ, Deziel DJ, Liau KH, Chen MF, Liu KH, Su CH, Chan ACW, Yoon DS, Choi IS, Jonas E, Chen XP, Fan ST, Ker CG, Gimenez ME, Kitano S, Inomata M, Mukai S, Higuchi R, Hirata K, Inui K, Sumiyama Y, Yamamoto M. Tokyo Guidelines 2018: antimicrobial therapy for acute cholangitis and cholecystitis. J Hepatobiliary Pancreat Sci. 2018 Jan;25(1):3-16. doi: 10.1002/jhbp.518. Epub 2018 Jan 9. PMID 29090866
- [Background] Gu XX, Zhang MP, Zhao YF, Huang GM. Clinical and microbiological characteristics of patients with biliary disease. World J Gastroenterol. 2020 Apr 14;26(14):1638-1646. doi: 10.3748/wjg.v26.i14.1638. PMID 32327912
- [Background] ASGE Standards of Practice Committee; Buxbaum JL, Abbas Fehmi SM, Sultan S, Fishman DS, Qumseya BJ, Cortessis VK, Schilperoort H, Kysh L, Matsuoka L, Yachimski P, Agrawal D, Gurudu SR, Jamil LH, Jue TL, Khashab MA, Law JK, Lee JK, Naveed M, Sawhney MS, Thosani N, Yang J, Wani SB. ASGE guideline on the role of endoscopy in the evaluation and management of choledocholithiasis. Gastrointest Endosc. 2019 Jun;89(6):1075-1105.e15. doi: 10.1016/j.gie.2018.10.001. Epub 2019 Apr 9. PMID 30979521
- [Background] Chandra S, Klair JS, Soota K, Livorsi DJ, Johlin FC. Endoscopic Retrograde Cholangio-Pancreatography-Obtained Bile Culture Can Guide Antibiotic Therapy in Acute Cholangitis. Dig Dis. 2019;37(2):155-160. doi: 10.1159/000493579. Epub 2018 Oct 3. PMID 30282078
- [Background] Negm AA, Schott A, Vonberg RP, Weismueller TJ, Schneider AS, Kubicka S, Strassburg CP, Manns MP, Suerbaum S, Wedemeyer J, Lankisch TO. Routine bile collection for microbiological analysis during cholangiography and its impact on the management of cholangitis. Gastrointest Endosc. 2010 Aug;72(2):284-91. doi: 10.1016/j.gie.2010.02.043. Epub 2010 Jun 11. PMID 20541201
- [Background] Hillenkamp F, Karas M, Beavis RC, Chait BT. Matrix-assisted laser desorption/ionization mass spectrometry of biopolymers. Anal Chem. 1991 Dec 15;63(24):1193A-1203A. doi: 10.1021/ac00024a002. No abstract available. PMID 1789447